CLINICAL TRIAL: NCT04690959
Title: Comparative Effects of Tensioning and Sliding Neural Mobilization on Nerve Root Function :Randomized Controlled Trial
Brief Title: Comparative Effects of Tensioning and Sliding Neural Mobilization on Nerve Root Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Associate professor-chair of Physiotherapy Department Affiliation: University of Sharjah, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USharjah 2021
Record Dates: First submitted 2020-12-26; First posted 2020-12-31 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Physical and Rehabilitation Medicine
Keywords: Randomized controlled trial; Neurodynamics; evoked potential; somatosensory

STUDY DESIGN:
Intervention Model Description: A prospective, parallel-group, randomized clinical trial participants will be randomly assigned to the control group or one of the 2 intervention groups. One group received neural gliding mobilization and the other neural tensioning mobilization, both targeting the median nerve
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants as well as The assessor, who took the measurements for both the intervention and control groups, was blinded to the subject's group, while the treating therapist was not blinded to the treatment intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neural gliding mobilization (Experimental): Initial participant positioning for gliding will be : lying in supine, shoulder at approximately 90 of abduction, wrist in neutral, elbow at 90 flexion and head/neck neutral. From this starting position, participants actively and simultaneously will perform extension of the elbow (to 45) and ipsilateral neck flexion (to approximately 45) and then returned to 90 of elbow flexion and 45 of contralateral neck flexion while maintaining the shoulder at 90 abduction. According to Silva et al., (2014) this combination of movements was the one that promoted the greatest excursion of the median nerve (10.2 mm) . For gliding, four series of 10 movements at a rhythm of approximately 6 s per cycle and 1-min rest between series was performed.
  Interventions: Other: neural mobilization
- Neural tensioning mobilization (Experimental): Tensioning will be performed with the subject lying supine. The investigator will perform the upper limb neurodynamic test as reported by Butler (2000): shoulder depression; 110 of shoulder abduction; external shoulder rotation; wrist and fingers extension; forearm supination and then elbow extension. The final test position will be defined as either i) end of joint amplitude or ii) the joint amplitude that provokes pain, paresthesia or numbness. In this case, a decrease of 5 to 10 of range of motion (elbow extension) will be allowed for symptoms to disappear and from this end position the investigator will perform repetitive movements of approximately 10 of elbow flexion/extension while maintaining the test end position for all the other joints. For tensioning, four series of 10 movements at a rhythm of approximately 6 s per cycle and 1-min rest between series will be performed. After each cycle of 10 repetitions, the position will be held for 10 seconds.
  Interventions: Other: neural mobilization
- Control (Sham Comparator): Participants in the sham group will receive a treatment consisting of maneuvers that mimic the neural mobilization treatment but not to stress the neural tissues in the upper extremity. The sham mobilization consists of passively positioning the participants in the following consecutive positions: (1) a neutral cervical spine (0° of lateral flexion), (2) 45°of shoulder abduction without scapula depression, and (3) 45° of shoulder external rotation combined with 45° of elbow flexion with forearm pronation. This will be immediately followed by 10 cycles of passive wrist flexion/extension at a rate of approximately 6 seconds per cycle (3 seconds into extension and 3 seconds into flexion) . Upon moving from wrist flexion to extension, an initial sense of resistance will be used as a sign to alternate directions. Following the 10th cycle, a static hold will be maintained while in wrist flexion for 10 seconds.
  Interventions: Other: Sham intervention

INTERVENTIONS:
Other: neural mobilization — Neural mobilization, or neurodynamics, is a movement-based intervention aimed at restoring the homeostasis in and around the nervous system.
  Other Names: neurodynamics
  Arms: Neural gliding mobilization; Neural tensioning mobilization
Other: Sham intervention — it is faked neural mobilization that mimic the neural mobilization treatment but believed not to stress the neural tissues in the upper extremity.
  Arms: Control

SUMMARY:
the current study will try to answer the question: Is it theoretically possible, that increased longitudinal stress on nerve root from sliding or tensioning intervention may subtly affect the neural function? Our hypothesis is that tensioning and sliding, differently affect the neural function.

DETAILED DESCRIPTION:
A prospective, parallel randomized, controlled study will be conducted at a research laboratory of our University. Participant recruitment will begin following approval from the Ethics Committee .The patients will participate in the study after signing an informed consent form prior to data collection.

Per inclusion criteria, subjects will be between 18 and 50 years of age, not currently experiencing any neck or dominant upper extremity symptoms, do not have a history significant for a chronic painful condition, and will not using pain relievers. Prior to participating in any study-related procedures, participants will read and signed an informed consent form approved by the Institutional Review Board.

Participants will be divided into three groups; One group will receive neural gliding mobilization and the other neural tensioning mobilization, both targeting the median nerve.

. the third group will receive sham neural mobilization intervention . Participants were not given information on which neural mobilization technique they were receiving; they were only told that they could receive one of two different neural mobilization techniques. Six sessions will be given every other day for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* not currently experiencing any neck or dominant upper extremity symptoms.
* do not have a history significant for a chronic painful condition.
* do not using pain relievers.

Exclusion Criteria:

* inflammatory joint disease or other systemic pathologies.
* prior history of overt injury and surgery relating to the musculoskeletal system.
* disorder related to the spine and extremities.
* musculoskeletal pain in the last three months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Change in dermatomal somatosensory evoked potentials | baseline (pre-treatment) , 2 weeks ,through study completion, an average of 1 week
  In all dermatomes, 2 complete recording runs will be undertaken during each session with averages of 250 to 1200 cortical responses from scalp surface recording electrodes (C3'-C4' in a 10-20 electrode configuration) of the contralateral scalp to the stimulated dermatomes being stimulated. The impedance of ground and scalp electrodes will be maintained at < 5 k Cutaneous areas of L3,L4,L5, S1 sensory roots will be stimulated in lower limb with the electrical impulses of 0.2 ms duration, frequency of 3.3 Hz and intensity 3 times higher than the sensory threshold will be determined individually for each subject.

SECONDARY OUTCOMES:
Change in Skin Sympathetic response | baseline (pre-treatment) , 2 weeks ,through study completion, an average of 1 week
  For measurement of the Skin Sympathetic response, electromyography equipment will be used. The skin temperature will be maintained at 32° )by making the stability of room temperature around 26° C, asking subjects to stay in the room for 20 minutes with that temperature before the examination and prevent local warm-up for extremities) . Active surface electrodes will be attached on the palmar side, and the references will be placed on the dorsum of the hand. The stimulus will be given at the wrist contralateral to the recording side. The latency and peak to peak amplitude will be determined. Sympathetic skin response will be considered absent if there is no response after ten stimuli.
Change in Pressure pain threshold | baseline (pre-treatment) , 2 weeks of treatment and at 1 week following the end of treatment
  An algometer will be used to measure Pressure pain threshold at both the thenar eminence and the proximal third of the right ventral forearm. . Before measurements on these points will be taken, Pressure pain threshold measurement will be demonstrated in the opposite upper limb to familiarize the patient with the procedure. Participants will be instructed to say "stop" when the sensation changed from pressure to pain. The Pressure pain threshold will be measured with the patient's hand and forearm in supination and supported on a table. Three measurements will be taken at each point. The mean value was used for between groups comparisons. A 30-second resting period will be allowed between each measurement. The pressure will be applied at a rate of 3 N/s up to a maximum of 60 N, which was not exceeded because of the risk of tissue damage.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Moustafa, associate professor, Principal Investigator — University of Sharjah
Locations (2):
- United Arab Emirates (2):
  - Ibrahim Moustafa, Sharjah city, United Arab Emirate
  - University of Sharjah, Sharjah city

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available to other researchers